CLINICAL TRIAL: NCT05389930
Title: Cannabis' Impact on Alcohol Consumption: Integrating Laboratory and Ecological Momentary Assessment Methods
Brief Title: Cannabis' Impact on Alcohol Consumption
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022003195; R01AA029711 (NIH)
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Drinking; Cannabis Use; Cannabis; Alcohol Use Disorder
Keywords: alcohol; cannabis; marijuana; addiction; cannabinoid; tetrahydrocannabinol; cannabidiol
MeSH Terms: conditions — Alcohol Drinking; Marijuana Abuse; Alcoholism; Behavior, Addictive | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Mixed factorial design will use a 3 (within-subjects; cannabinoid dose: 9.53% THC/0.06% CBD, 11.27% CBD/0.35% THC, placebo) X 2 (between-subjects; cannabis + an alcohol-priming dose (0.3 g/kg) versus cannabis + alcohol placebo)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are masked. Outcome assessors who have contact with participants are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- THC-dominant cannabis dose (Experimental): 367 mg of cannabis plant material with 9.53% THC and 0.09% CBD and 217 mg of placebo cannabis plant material will be mixed and smoked in a handheld pipe
  Interventions: Drug: Alcohol; Drug: Alcohol placebo
- CBD-dominant cannabis dose (Experimental): 367 mg of cannabis plant material with 11.27% CBD and 0.35% THC and 217 mg of placebo cannabis plant material will be mixed and smoked in a handheld pipe
  Interventions: Drug: Alcohol; Drug: Alcohol placebo
- Placebo (Placebo Comparator): 584 mg of cannabis plant material will be smoked in a handheld pipe
  Interventions: Drug: Alcohol; Drug: Alcohol placebo
- Alcohol priming dose (Experimental): Alcohol: 0.3 g/kg. Alcohol priming drink is designed to raise blood alcohol levels to 0.03 g/dl and be consumed in 5 minutes. The drink is mixed using 80-proof liquor and juice. Participants are randomized to receive either the experimental alcohol priming dose or alcohol placebo.
  Interventions: Drug: THC-dominant cannabis; Drug: CBD-dominant cannabis; Drug: Cannabis placebo
- Alcohol placebo dose (Placebo Comparator): Placebo beverage contains only juice and a negligible trace of alcohol for masking. The weight and sex-adjusted volume of alcohol and non-alcohol containing beverages will be equal. Participants are randomized to receive either the experimental alcohol priming dose or alcohol placebo.
  Interventions: Drug: THC-dominant cannabis; Drug: CBD-dominant cannabis; Drug: Cannabis placebo

INTERVENTIONS:
Drug: THC-dominant cannabis — Smoked cannabis with 9.53% THC and 0.09% CBD
  Arms: Alcohol placebo dose; Alcohol priming dose
Drug: CBD-dominant cannabis — Smoked cannabis with 0.35% THC and 11.27% CBD
  Arms: Alcohol placebo dose; Alcohol priming dose
Drug: Cannabis placebo — Smoked placebo cannabis plant material
  Arms: Alcohol placebo dose; Alcohol priming dose
Drug: Alcohol — Drink containing 0.3 g/kg of alcohol
  Arms: CBD-dominant cannabis dose; Placebo; THC-dominant cannabis dose
Drug: Alcohol placebo — Placebo beverage contains only juice and a negligible trace of alcohol for masking
  Arms: CBD-dominant cannabis dose; Placebo; THC-dominant cannabis dose

SUMMARY:
This study employs a repeated measures experimental design to examine the effect of THC-dominant dose of cannabis and CBD-dominant dose of cannabis, relative to placebo, on subsequent drinking in an alcohol choice task in which participants choose either to drink or receive monetary reinforcement for drinks not consumed. Cannabis will be administered simultaneously with an alcohol-priming dose or alcohol placebo.

The study will enroll up to 350 nontreatment-seeking heavy episodic alcohol drinkers who use cannabis weekly.

DETAILED DESCRIPTION:
This study employs a repeated measures experimental design to examine the effect of THC-dominant (9.53% THC and 0.09% CBD) dose of cannabis and CBD-dominant (0.35% THC and 11.27% CBD) dose of cannabis, relative to placebo, on subsequent drinking in an alcohol choice task in which participants choose either to drink or receive monetary reinforcement for drinks not consumed. Cannabis will be administered simultaneously with an alcohol-priming dose or alcohol placebo. The study will enroll up to 350 nontreatment-seeking heavy episodic alcohol drinkers who use cannabis weekly to obtain the final sample of 200 with complete data. Participants will be tested at a baseline session, during three experimental sessions, and then during a subsequent 4-week period in the natural environment using a smart-phone application. Findings have important implications for cannabis regulatory science and alcohol use disorder treatment by addressing the relative impact of specific cannabinoids as well as contextual risk in cannabis-alcohol co-use.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 50
* English-speaking
* cannabis smoking in past two months
* heavy drinking in past two months
* in good physical health and weighing < 250 lbs
* zero breath alcohol at each visit

Exclusion Criteria:

* positive pregnancy test
* nursing
* positive urine toxicology screen for drugs other than cannabis
* interest to quit or receive treatment for cannabis or alcohol use

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
ml of alcohol consumed | post-smoking during two-hours of the alcohol choice task
  ml of alcohol consumed during the alcohol choice task

CONTACTS AND LOCATIONS:
Overall Officials: Jane Metrik, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States